CLINICAL TRIAL: NCT05704530
Title: Personalized Multimodal Treatment for Resectable Esophageal Cancer by Detecting Minimal Residual Disease Using Circulating Tumor DNA: a Multicentric Prospective Study
Brief Title: Liquid Biopsies in Esophageal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Kom Op Tegen Kanker (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: S67328
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Three distinct patient groups are defined, depending on the therapeutic scenario patients undertake. Patient management is standard of care. No investigational medicinal product (IMP) is involved.
  Trial is considered low interventional due to addition of extra blood samples, otherwise would be observational.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1. primary resection then follow-up (Other): Scenario 1: primary resection then follow-up - Study-specific liquid biopsies will be collected in 98 patients, at the time of routine labs. Samples will be acquired before resection, at 6-8 weeks, 6 and 12 months after resection.
  Interventions: Other: Blood sample
- 2. chemoradiation followed by resection and follow-up (Other): Scenario 2: chemoradiation followed by resection and follow-up - Study-specific liquid biopsies will be collected in 50 patients. Samples will be acquired before the start of chemoradiation, before surgery, 6-8 weeks, 6 and 12 months after surgery. A subgroup of patients will undertake adjuvant immunotherapy and will constitute Group 3. Timing of sampling will be adjusted accordingly as per study flowcharts.
  Interventions: Other: Blood sample
- 3. chemoradiation followed by resection followed by adjuvant immunotherapy (Other): chemoradiation followed by resection followed by adjuvant immunotherapy - Study-specific liquid biopsies will be collected in 100 patients. Samples will be acquired before the start of chemoradiation, before surgery, 6-8 weeks after surgery and during adjuvant immunotherapy every 3 months including a sample at the end of treatment.
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Retrospective collection of leftover tissue from standard of care biopsies or resection specimens and prospective collection of additional blood samples for study-specific analyses at specific timepoints, at the same time as routine labs are foreseen. No additional venipunctures are expected.

SUMMARY:
Purpose of this study is to determine the value of liquid biopsies, e.g. testing of minimal residual disease (MRD) by using liquid biopsies to measure circulating tumour DNA (ctDNA) at diagnosis and during the multimodal and multidisciplinary curative-intent treatment of resectable esophageal cancer.

DETAILED DESCRIPTION:
Multicentric, retrospective and prospective components.

Retrospective collection of leftover tissue from standard of care biopsies or resection specimens and prospective collection of additional blood samples for study-specific analyses at specific timepoints, at the same time as routine labs are foreseen. No additional venipunctures are expected.

Three distinct patient groups are defined, depending on the therapeutic scenario patients undertake:

Scenario 1: primary resection then follow-up - Study-specific liquid biopsies will be collected in 98 patients, at the time of routine labs. Samples will be acquired before resection, at 6-8 weeks, 6 and 12 months after resection.

Scenario 2: chemoradiation followed by resection and follow-up - Study-specific liquid biopsies will be collected in 50 patients. Samples will be acquired before the start of chemoradiation, before surgery, 6-8 weeks, 6 and 12 months after surgery. A subgroup of patients will undertake adjuvant immunotherapy and will constitute Group 3. Timing of sampling will be adjusted accordingly as per study flowcharts.

Scenario 3: chemoradiation followed by resection followed by adjuvant immunotherapy - Study-specific liquid biopsies will be collected in 100 patients. Samples will be acquired before the start of chemoradiation, before surgery, 6-8 weeks after surgery and during adjuvant immunotherapy every 3 months including a sample at the end of treatment.

Patient management is standard of care. No investigational medicinal product (IMP) is involved.

Specific clinicopathological variables will be collected in a RedCap electronic Case Report Form and analysed as per statistical analysis plan.

ELIGIBILITY:
Key inclusion criteria are:

1. Male or female, age > 18 years
2. New diagnosis of esophageal cancer, pathologically confirmed squamous cell carcinoma (ESCC) or adenocarcinoma (EAC)
3. Clinically staged - cT1-4 N0-2 M0 (local or locally advanced, resectable)
4. Eligible for multidisciplinary treatment as assessed by MDT
5. Able to provide informed consent (ICF) according to Good Clinical Practice and national/European regulations

Key exclusion criteria are:

1. (Oligo)metastatic disease
2. Histologically or cytologically confirmed diagnosis other than squamous cell carcinoma or adenocarcinoma (eg. neuroendocrine carcinoma, lymphoma…)
3. Other active malignancies
4. Previous exposure to chemoradiation (prior to MDT)
5. Treatment plan after MDT: neoadjuvant chemotherapy with no radiation or chemoradiation with definitive intent (surgery is not planned)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Estimated)
Dates: Start 2023-03-29 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess the potency of ctDNA MRD variant allele frequency to improve clinical staging at diagnosis of esophageal cancer. | 12 months
  To assess whether ctDNA concentration can significantly contribute to preoperative staging in esophageal cancer, to define a significant cut-off value of ctDNA concentration with optimal sensitivity and specificity and validate the results.
To correlate the presence of minimal residual disease after resection as assessed by ctDNA with disease recurrence. | 12 months
  To compare the two groups ctDNA positive and negative post-resection in terms of progression-free survival and overall survival (Kaplan-Meier time-to-event) and evaluate the performance of ctDNA to predict disease recurrence (Cox proportional hazards model).
To observe the ctDNA MRD dynamics during adjuvant immunotherapy . | 12 months
  To describe the dynamics of ctDNA concentration (proportion of clearance of positive ctDNA) during standard of care adjuvant immunotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Dekervel, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (4):
- Belgium (4):
  - UZA, Antwerp
  - UZ Gent, Ghent
  - UZLeuven, Leuven
  - AZ Delta, Roeselare

IPD SHARING:
Plan to Share IPD: No